CLINICAL TRIAL: NCT01762839
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Design, Study With an Open-Label Positive-Control, to Assess the Cardiac Safety of Oritavancin in Healthy Volunteers
Brief Title: A Study to Assess the Cardiac Safety of Oritavancin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDCO-ORI-12-02
Record Dates: First submitted 2012-12-12; First posted 2013-01-08 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oritavancin (Experimental): Single-dose intravenous (IV) oritavancin diphosphate
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate
- Placebo (Placebo Comparator): Single-dose IV placebo
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Moxifloxacin tablet
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Single-Dose IV Oritavancin Diphosphate — Intravenous oritavancin was administered via 2 dedicated, peripheral venous lines, 1 in each arm. The infusion lasted approximately 3 hours.
  Other Names: Oritavancin Diphosphate
  Arms: Oritavancin
Drug: Placebo — Intravenous placebo was administered via 2 dedicated, peripheral venous lines, 1 in each arm. The infusion lasted approximately 3 hours.
  Arms: Placebo
Drug: Moxifloxacin — Participants randomized to the open-label moxifloxacin treatment arm only received a 400-mg moxifloxacin tablet and did not receive a placebo infusion.
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of the study was to generate cardiac safety data using a supratherapeutic oritavancin dose of 1600 milligrams (mg).

DETAILED DESCRIPTION:
This study was a single-center, double-blind, randomized, placebo-controlled, parallel-design study with an open-label, positive-control moxifloxacin arm to evaluate the effect of supratherapeutic dose of oritavancin on the QT and QT corrected for pulse rate (QTc) intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent before initiation of any study related procedures and willing to comply with all required study procedures.
2. Healthy, male and female between 18 and 60 years old, body mass index between 18 and 30 kilograms/meter squared.
3. In good health based upon results of medical history, physical examination, no clinically significant 12-lead electrocardiogram (ECG) results, and laboratory test results.
4. Serum magnesium and potassium levels within the normal range at Screening.
5. Agreed to abstain from alcohol, caffeine-, and xanthine-containing products, all kind of energy drinks and the consumption of grapefruit juice and orange juice from 48 hours before study drug administration until completion of the follow-up visit.

Exclusion Criteria:

1. History of immune-related hypersensitivity reaction to glycopeptides (such as vancomycin, televancin, daptomycin, or teicoplanin) or any of their excipients. Note: participants who had histamine-like infusion reactions to a glycopeptide were not excluded.
2. A resting pulse rate < 50 beats per minute (bpm) or > 100 bpm.
3. Systolic blood pressure < 90 millimeters of mercury (mmHg) or diastolic blood pressure < 50 mmHg.
4. A QTc with the Fridericia correction > 450 microseconds (msec) (males) or > 470 msec (females).
5. Respiratory difficulties, or a history of asthma or chronic obstructive pulmonary disease.
6. Use of any prescription drug or over-the-counter medications or herbal preparations within 14 days or 5-times the elimination half-life (whichever was longer) prior to starting the study (except for acetaminophen; birth control pills; implantable or injectable birth control; and estrogen, testosterone, and/or progesterone replacement in menopausal women).
7. Unwilling to abstain from smoking for the duration of the study.
8. Any clinically significant, underlying abnormalities in rhythm, conduction, or morphology of the resting ECG that may have interfered with the interpretation of QTc interval changes.
9. Positive result for the urine or serum human chorionic gonadotropin test administered at Screening (females with childbearing potential).
10. A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents, or siblings) of either a long or a short QT syndrome.
11. Personal history of unexplained syncope.
12. Women who were pregnant or nursing, or who were of childbearing potential and unwilling to use at least 2 acceptable methods of birth control (for example, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier method(s) or male partner sterilization). Women ≥ 2 years postmenopausal or surgically sterile were exempt from this exclusion.
13. A history of hypersensitivity to moxifloxacin or any member of the quinolone class of antimicrobial agents.
14. Positive virology screen for human immunodeficiency virus or hepatitis B or C virus, respectively.
15. Participated in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment.
16. Any condition, which in the opinion of the Investigator would put the participant at increased risk from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-12-27 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-02-11 (Actual)

PRIMARY OUTCOMES:
Placebo-adjusted change from Baseline in QTcF | predose, 3,3.5,4,5,6,7,9,11,15,24 hours post infusion start time
  Placebo-adjusted change from baseline in QTcF (QTc with the Fridericia correction) between each treatment and placebo.

SECONDARY OUTCOMES:
Placebo-adjusted change from baseline in QTcB, HR, RR, PR, and QRS interval analyses. | predose, 3,3.5,4,5,6,7,9,11,15,24 hours post infusion start time
  Placebo-adjusted change from baseline in QTcB, HR, RR, PR, and QRS interval analyses.
Placebo adjusted change from Baseline in the appearance or worsening of ST, T and U-wave morphology. | predose, 3,3.5,4,5,6,7,9,11,15,24 hours post infusion start time
  Placebo adjusted change from baseline in the appearance or worsening of ST, T and U-wave morphology.
Effects on the QTc interval related to plasma concentration levels of oritavancin | predose, 3,3.5,4,5,6,7,9,11,15,24 hours post infusion start time
  Compare the effects on the QTc interval to the plasma levels of oritavancin using concentration-effect modeling
Evaluate the number of volunteers with adverse events or abnormalities in lab/urine results and safety ECGs as measures of safety and tolerability | Day 0 through Day 7
  Compare safety and tolerability in healthy volunteers after a single IV dose of 1600 mg oritavancin

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States